CLINICAL TRIAL: NCT06628791
Title: Effects of Oral Intake of BK329 on Body Fat Reduction in Adults With Overweight or Obesity: a Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: BK329 and Body Fat Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Sang Yeoup Lee, Professor, MD, PhD, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 12-2023-002
Record Dates: First submitted 2024-10-04; First posted 2024-10-08 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Obesity and Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BK329 group (Experimental): This group takes BK329 for 12 weeks.
  Interventions: Dietary Supplement: BK329
- Placebo group (Placebo Comparator): This group takes placebo for 12 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: BK329 — Lactococcus lactics. subsp. lactis CAB701(KCCM13360P) 400 mg/day for 12 weeks
  Arms: BK329 group
Dietary Supplement: Placebo — Placebo 400 mg/day for 12 weeks
  Arms: Placebo group

SUMMARY:
This clinical trial aims to determine whether BK329 reduces body fat in adults with overweight or obesity and to assess its safety.

The main questions are:

* Does BK329 reduce body fat in participants?
* What side effects occur when participants take BK329?

DETAILED DESCRIPTION:
Researchers will compare BK329 to a placebo to evaluate its effectiveness in reducing body fat.

Participants will:

* Take BK329 or a placebo daily for 12 weeks.
* Visit the clinic every six weeks for checkups and tests.

ELIGIBILITY:
Inclusion Criteria:

* individuals with a Body Mass Index (BMI) between 23 and 30 kg/m2.
* Individuals who have provided written consent on the consent form.

Exclusion Criteria:

* Subjects with severe cerebrovascular disease (e.g., stroke, cerebral hemorrhage), heart disease (e.g., angina, myocardial infarction, heart failure, arrhythmia requiring treatment), or malignant tumors within the last 6 months. (However, subjects with a history of these diseases who are clinically stable may participate at the investigator's discretion.)
* Uncontrolled hypertensive patients (blood pressure ≥160/100mmHg, measured after 10 minutes of rest).
* Diabetic patients with poor blood glucose control (fasting glucose ≥160mg/dL).
* Subjects undergoing treatment for hypothyroidism or hyperthyroidism.
* Subjects with creatinine levels ≥ 2 times the upper limit of the research institution's normal range.
* Subjects with aspartate transaminase or alanine transaminase levels ≥ 3 times the upper limit of the research institution's normal range.
* Subjects experiencing severe gastrointestinal symptoms such as heartburn or indigestion (lactose intolerance).
* Subjects who have taken weight-altering drugs (absorption inhibitors, appetite suppressants, obesity-related supplements, psychiatric drugs, beta-blockers, diuretics, contraceptives, steroids, or female hormones) within the last month.
* Subjects who have participated in commercial weight loss programs within the last 3 months.
* Subjects who have participated in or plan to participate in another clinical trial within the last month.
* Alcohol abusers.
* Subjects who quit smoking within the last 3 months.
* Pregnant or breastfeeding women or those planning pregnancy during the trial period.
* Subjects with allergies to any components of the study foods.
* Subjects deemed inappropriate for the study by the investigator for other reasons.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-01-26 (Actual); Primary Completion 2024-07-08 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Total body fat (kg) | 12 weeks
  Using dual-energy X-ray absorptiometry at baseline and 12 weeks

SECONDARY OUTCOMES:
Body fat percentage | 12 weeks
  Using dual-energy X-ray absorptiometry at baseline and 12 weeks
Lean body mass (kg) | 12 weeks
  Using dual-energy X-ray absorptiometry at baseline and 12 weeks
Body mass index (kg/m2) | 12 weeks
  Measured at baseline and 12 weeks
Body weight (kg) | 12 weeks
  Measured at baseline and 12 weeks
Waist-to-hip ratio | 12 weeks
  Measured at baseline and 12 weeks
Total cholesterol level (mg/dl) | 12 weeks
  Measured at baseline and 12 weeks
Triglycerides level (mg/dL) | 12 weeks
  Measured at baseline and 12 weeks
High-density lipoprotein cholesterol levels (mg/dL) | 12 weeks
  Measured at baseline and 12 weeks
Low-density lipoprotein cholesterol levels (mg/dL) | 12 weeks
  Measured at baseline and 12 weeks
Free fatty acid level (mg/dL) | 12 weeks
  Measured at baseline and 12 weeks
High-sensitivity C-reactive protein (mg/dL) | 12 weeks
  Measured at baseline and 12 weeks
Total immunoglobulin E level (IU/mL) | 12 weeks
  Measured at baseline and 12 weeks
Neutrophil-to-lymphocyte ratio | 12 weeks
  Measured at baseline and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sang Yeoup Lee, MD, PhD, Principal Investigator — Pusan National University Yangsan Hospital
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, South Korea

IPD SHARING:
Plan to Share IPD: No